CLINICAL TRIAL: NCT06870006
Title: Psychotropic-Drug-induced QT Prolongation and ECG Monitoring in the Pediatric Population
Status: Recruiting | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: PDP-QT
Record Dates: First submitted 2025-02-27; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Eating Disorders; Mood Disorders in Children and Adolescents; Psychotic Disorder; QTc Intervals Changes
Keywords: QTc interval; psychotropic drugs
MeSH Terms: conditions — Feeding and Eating Disorders; Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Monotherapy: Patients taking only one drug acting on QT interval
- Monotherapy to monotherapy: Patients who have switched from a drug acting on QT interval to another
- Polytherapy: Patients taking more than one drug acting on QT interval

SUMMARY:
Electrocardiogram (ECG) Q-T prolongation is a cardiac electrophysiological disorder associated with the occurrence of arrhythmias potentially fatal. Several psychotropic drugs are associated with an increased risk of QT prolongation, which is why in clinical practice a baseline ECG is performed before a psychotropic drug is prescribed. However, there are no validated protocols establishing when to repeat this examination or describing clinical events when this examination should be repeated in clinical follow-up.

The study aims to investigate the incidence of QTc prolongation events as a side effect of chronic psychotropic drug administration. For this purpose, ECGs will be recorded and confounding factors of patients at the beginning of psychotropic therapy and after 3, 6 and 12 months will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to psychiatry ward
* Starting a psychotropic drug acting on QT interval

Exclusion Criteria:

* Age >18aa
* History of administration of drug acting on QT interval in the 3 months prior

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents referring to psychiatry services in one the participating hospitals starting a new prescription for a psychotropic drug acting on QT interval.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Changes in QT interval | Baseline, 1, 3, 6, 12, 18 months post- enrollment

SECONDARY OUTCOMES:
Number of Cardiac events | Baseline, 1, 3, 6, 12, 18 months post- enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Meyer IRCCS, Florence, FI, Italy

IPD SHARING:
Plan to Share IPD: Undecided